CLINICAL TRIAL: NCT00009737
Title: An Open-Label Randomized Phase III Study Comparing Xeloda (Capecitabine) With IV Bolus 5-Fluorouracil in Combination With Low-Dose Leucovorin as Adjuvant Chemotherapy in Patients Who Underwent Surgery for Dukes C Colon Cancer
Brief Title: A Study of Xeloda (Capecitabine) Compared With 5-Fluorouracil in Combination With Low-Dose Leucovorin in Patients Who Have Undergone Surgery for Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M66001
Record Dates: First submitted 2001-02-02; First posted 2004-03-17 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Capecitabine

ARMS (2):
- Capecitabine (Experimental): Participants received capecitabine 1250 milligram per square meter (mg/m ^ 2) orally, twice a day, for 14 days, followed by a 7-day rest period without treatment, as an intermittent therapy in a 3-week cycle for 8 cycles (24 weeks).
  Interventions: Drug: Capecitabine [Xeloda]
- 5-Fluorouracil + Leucovorin (Active Comparator): Participants received leucovorin 20 mg/m ^ 2 followed by 5-fluorouracil at 425 mg/m ^ 2, by rapid intravenous injection, daily, from Days 1 to 5 of the first week in each 4-week cycle for 6 cycles (24 weeks).
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: 5-Fluorouracil — 425mg/m2 iv daily from day 1 to day 5 every 28 days.
  Arms: 5-Fluorouracil + Leucovorin
Drug: Leucovorin — 20mg/m2 iv daily from day 1 to day 5 every 28 days.
  Arms: 5-Fluorouracil + Leucovorin
Drug: Capecitabine [Xeloda] — 1250mg/m2 po bid on days 1-14 every 21 days.
  Arms: Capecitabine

SUMMARY:
This 2 arm study will compare the safety and efficacy of oral Xeloda, or 5-fluorouracil in combination with leucovorin, in patients who have undergone surgery for colon cancer. Patients will be randomized to receive either Xeloda 1250mg/m2 po bid on days 1-14 every 21 days, or leucovorin 20mg/m2 iv + 5-fluorouracil 425mg/m2 iv daily from day 1 to day 5 every 28 days. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-75 years of age;
* histologically confirmed colon cancer with potentially curative resection of the tumor within 8 weeks before study initiation.

Exclusion Criteria:

* previous chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1987 (Actual)
Dates: Start 1998-11; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (115):
- United States (17):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Fountain Valley, California
  - Los Angeles, California
  - Hartford, Connecticut
  - Miami, Florida
  - Decatur, Georgia
  - Columbia, Missouri
  - St Louis, Missouri
  - Albany, New York
  - Buffalo, New York
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Tyler, Texas
  - Seattle, Washington
- Buenos Aires, Argentina
- Australia (11):
  - Adelaide
  - Bendigo
  - Brisbane
  - Fitzroy
  - Kurralta Park
  - Melbourne
  - Perth
  - Port Macquarie
  - St Leonards
  - Sydney
  - Wodonga
- Austria (7):
  - Hall in Tirol
  - Innsbruck
  - Klagenfurt
  - Linz
  - Oberwart
  - Sankt Pölten
  - Vienna
- Brussels, Belgium
- Brazil (4):
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
  - Sorocaba
- Canada (6):
  - Calgary, Alberta
  - Kelowna, British Columbia
  - Winnipeg, Manitoba
  - Ottawa, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
- Germany (16):
  - Berlin
  - Braunschweig
  - Freiburg im Breisgau
  - Göttingen
  - Grenzach-Wyhlen
  - Halle
  - Hanover
  - Kassel
  - Lehrte
  - Magdeburg
  - München
  - Oldenburg
  - Ravensburg
  - Regensburg
  - Villingen-Schwenningen
  - Wuppertal
- Israel (4):
  - Haifa
  - Petah Tikva
  - Rehovot
  - Tel Aviv
- Italy (18):
  - Aviano
  - Bergamo
  - Bologna
  - Cuneo
  - Genova
  - Livorno
  - Mantova
  - Milan
  - Mirano
  - Modena
  - Napoli
  - Pisa
  - Roma
  - Terni
  - Torino
  - Vecchiazzano
  - Venezia
  - Vicenza
- Portugal (2):
  - Lisbon
  - Porto
- Spain (9):
  - Bilbao
  - Córdoba
  - El Palmar Murcia
  - Elche
  - Jaén
  - Madrid
  - Navarra
  - Palma de Mallorca
  - Valencia
- Switzerland (5):
  - Basel
  - Bellinzona
  - Bern
  - Sankt Gallen
  - Zurich
- United Kingdom (14):
  - Aberdeen
  - Belfast
  - Cardiff
  - Edinburgh
  - Glasgow
  - Guildford
  - Leicester
  - Luton
  - Manchester
  - Newcastle upon Tyne
  - Northwood
  - Plymouth
  - Salisbury
  - Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1987 participants were recruited into the study across 164 centers in 25 countries. This study was conducted from 12 Nov 1998 to 01 Apr 2004.
Period: Overall Study
Arm/Group | Capecitabine | 5-Fluorouracil + Leucovorin
Started | 1004 | 983
Completed | 834 | 860
Not Completed | 170 | 123
Not completed — Adverse Event | 112 | 75
Not completed — Death | 4 | 6
Not completed — Lack of Efficacy | 17 | 15
Not completed — Violation of Selection Criteria at Entry | 13 | 9
Not completed — Other Protocol Violation | 1 | 0
Not completed — Refused Treatment | 15 | 16
Not completed — Lost to Follow-up | 1 | 1
Not completed — Administrative/Other Reasons | 7 | 1

BASELINE CHARACTERISTICS:
Population: All randomized population included all participants who were randomized to one of the two treatment arms, regardless of whether they received any study medication.
Groups:
- Capecitabine: Participants received capecitabine 1250 (mg/m ^ 2) orally, twice a day, for 14 days, followed by a 7-day rest period without treatment, as an intermittent therapy in a 3-week cycle for 8 cycles (24 weeks).
- Total: Total of all reporting groups
Arm/Group | Capecitabine | 5-Fluorouracil + Leucovorin | Total
Number analyzed (Participants) | 1004 | 983 | 1987
Age, Continuous [Median (Full Range); unit: Years] — For median age, summary is based on n=1985
  Years | 62.0 [25 to 80] | 63.0 [22 to 82] | 62.0 [22 to 82]
Sex/Gender, Customized [Number; unit: Participants]
  Female | 461 | 451 | 912
  Male | 542 | 532 | 1074
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Participants with disease-free survival were reported. Disease-free survival was assessed as the number of days between randomization and the first time at which relapse, a new occurrence of colon cancer, or death was recorded, or the last time at which a participant was known to be disease free (censoring time).
Time Frame: Approximately 3 years
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Capecitabine | 5-Fluorouracil + Leucovorin
Number analyzed (Participants) | 1004 | 983
Participants | 656 | 603
Statistical Analysis 1: Comparison: Capecitabine vs 5-Fluorouracil + Leucovorin; Test type: Non-Inferiority or Equivalence — Non-inferiority was tested by comparing the upper limit of the 95% confidence interval for the hazard ratio to the non-inferiority margin of 1.25 in a first step, and then of 1.20 in a second step; p = 0.053, Wald Chi-Square Test — For difference between arms, < 0.001 for non-inferiority; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.75 to 1.00]

2. Secondary Outcome: Relapse-Free Survival
Description: Participants with relapse-free survival were reported. Relapse-free survival was assessed as the number of days between randomization and the first time at which relapse, a new occurrence of colon cancer, or death was recorded, or the last time at which a participants was known to be disease free (censoring time), excluding deaths that were not related to treatment or to disease progression.
Time Frame: Approximately 3 years
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Capecitabine | 5-Fluorouracil + Leucovorin
Number analyzed (Participants) | 1004 | 983
Participants | 677 | 621
Statistical Analysis 1: Comparison: Capecitabine vs 5-Fluorouracil + Leucovorin; Test type: Non-Inferiority or Equivalence — Non-inferiority was tested by comparing the upper limit of the 95% confidence interval for the hazard ratio to the non-inferiority margin of 1.25; p = 0.041, Wald Chi-Square Test — For difference between arms, < 0.001 for non-inferiority; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.74 to 0.99]

3. Secondary Outcome: Overall Survival
Description: Participants with overall survival were reported. Overall survival was assessed as the number of days between randomization and death or the last time at which a participant was known to be alive (censoring time).
Time Frame: Approximately 3 years
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Capecitabine | 5-Fluorouracil + Leucovorin
Number analyzed (Participants) | 1004 | 983
Participants | 804 | 756
Statistical Analysis 1: Comparison: Capecitabine vs 5-Fluorouracil + Leucovorin; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.071, Wald Chi-Square Test — For difference between arms, < 0.001 for non-inferiority; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.69 to 1.01]

4. Secondary Outcome: Mean Change From Baseline in Global Health Status at Week 25
Description: Global health status was assessed as a sub scale of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30. It was scored on a scale of 0-100; where higher score indicates better quality of life. Wherever the scores for the participants were not available, the last value carried forward (LVCF) were used.
Time Frame: Baseline (Days -7 to 1) and at Week 25
Population: The safety population included all participants who received at least one dose of capecitabine, 5-fluorouracil, or leucovorin and had at least one post baseline safety assessment (adverse events, laboratory test results, or vital signs).
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Capecitabine | 5-Fluorouracil + Leucovorin
Number analyzed (Participants) | 836 | 769
Score on a scale | 2.1 (0.80) | 2.6 (0.78)

5. Secondary Outcome: Number of Participants With Abnormalities for Blood Chemistry and Hematological Parameters
Description: Laboratory abnormalities were categorized according to the National Cancer Institute of Canada Common Toxicity Criteria (NCIC - CTC) grading system (May 1991 revised) as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (life- threatening). Participants with abnormalities in hemoglobin, granulocytes, lymphocytes, neutrophils, neutrophils/granulocytes, platelets, white blood cell, potassium, serum creatinine, sodium, total bilirubin, alanine transaminase, aspartate aminotransferase, alkaline phosphatase, calcium (hyper), and calcium (hypo) with Grades 1-4 were presented.
Time Frame: Up to Week 25
Population: The safety population comprises all participants who received at least one dose of capecitabine, 5-fluorouracil, or leucovorin and had at least one post baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Capecitabine | 5-Fluorouracil + Leucovorin
Number analyzed (Participants) | 995 | 974
Participants
  Alanine transaminase | 327 | 333
  Aspartate aminotransferase | 300 | 288
  Alkaline Phosphatase | 334 | 289
  Calcium (Hyper) | 67 | 68
  Calcium (Hypo) | 150 | 112
  Granulocytes | 20 | 43
  Hemoglobin | 691 | 650
  Lymphocytes | 778 | 744
  Neutrophils | 308 | 596
  Neutrophils/Granulocytes | 316 | 612
  Platelets | 182 | 160
  Potassium | 209 | 156
  Serum Creatinine | 157 | 138
  Sodium | 189 | 184
  Total Bilirubin | 501 | 185
  White blood cell | 220 | 409

6. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An Serious Adverse Events (SAEs) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Up to Week 29
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Capecitabine | 5-Fluorouracil + Leucovorin
Number analyzed (Participants) | 995 | 974
Participants
  All adverse events | 910 | 885
  Serious adverse events | 181 | 182

ADVERSE EVENTS:
Time Frame: Up to Week 29
Description: Adverse event is reported for safety population which consist of all participants who received at least one dose of capecitabine, 5-fluorouracil, or leucovorin and had at least one post baseline safety assessment.
Arm/Group | Capecitabine | 5-Fluorouracil + Leucovorin
Serious Adverse Events (participants affected / at risk) | 181/995 | 182/974
Other Adverse Events (participants affected / at risk) | 838/995 | 847/974
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=995) | 5-Fluorouracil + Leucovorin (N=974)
Diarrhoea (Gastrointestinal disorders) | 58 | 34
*Stomatitis all (Gastrointestinal disorders) | 4 | 25 — *Monthly Incidence of Hospitalization = (Number of Hospitalizations / (Days on Treatment + 28)) * 30.5
Abdominal pain (Gastrointestinal disorders) | 9 | 10
Small intestinal obstruction (Gastrointestinal disorders) | 7 | 10
Intestinal obstruction (Gastrointestinal disorders) | 9 | 3
Vomiting (Gastrointestinal disorders) | 5 | 7
Enteritis (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Subileus (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 2 | 1
Ileus paralytic (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 3
Colonic polyp (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Mechanical ileus (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Peritonitis (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal mucositis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 4
Neutropenic sepsis (Infections and infestations) | 0 | 5
Pneumonia (Infections and infestations) | 2 | 3
Abdominal abscess (Infections and infestations) | 2 | 1
Bronchopneumonia (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 0 | 3
Catheter related infection (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 0 | 2
Localised infection (Infections and infestations) | 2 | 0
Orchitis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1
Clostridium colitis (Infections and infestations) | 1 | 0
Fallopian tube abscess (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Incision site abscess (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Lower respiratory tract Infection (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Peritoneal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 17
Neutropenia (Blood and lymphatic system disorders) | 3 | 7
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 10 | 6
Thrombophlebitis (Vascular disorders) | 1 | 2
Thrombosis (Vascular disorders) | 2 | 1
Aortic aneurysm (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 2
Phlebitis (Vascular disorders) | 2 | 0
Phlebothrombosis (Vascular disorders) | 2 | 0
Thrombophlebitis superficial (Vascular disorders) | 2 | 0
Arteriopathic disease (Vascular disorders) | 0 | 1
Gangrene (Vascular disorders) | 0 | 1
Iliac vein thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemopneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 2
Angina pectoris (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Torsade de pointes (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 6 — General Disorders and Administration Site Conditions
Fatigue (General disorders) | 1 | 1 — General Disorders and Administration Site Conditions
Lethargy (General disorders) | 2 | 0 — General Disorders and Administration Site Conditions
Non-cardiac chest pain (General disorders) | 2 | 0 — General Disorders and Administration Site Conditions
Asthenia (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions
Chest pain (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions
Death (General disorders) | 0 | 1 — General Disorders and Administration Site Conditions
Malaise (General disorders) | 1 | 0 — General Disorders and Administration Site Conditions
Oedema peripheral (General disorders) | 0 | 1 — General Disorders and Administration Site Conditions
Rigors (General disorders) | 0 | 1 — General Disorders and Administration Site Conditions
Dehydration (Metabolism and nutrition disorders) | 8 | 7
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Ataxia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Cerebral artery occlusion (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0
Petit mal epilepsy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Anticonvulsant toxicity (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Intestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 2
Renal colic (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal insufficiency (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Palmar - plantar (Skin and subcutaneous tissue disorders) | 4 | 0
Erythrodysaesthesia syndrome Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin inflammation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
International normalised ratio Increased (Investigations) | 1 | 1
Blood triglycerides increased (Investigations) | 1 | 0
Blood urine (Investigations) | 1 | 0
Chest x-ray abnormal (Investigations) | 0 | 1
Tumour marker increased (Investigations) | 0 | 1
Anaphylactoid reaction (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 1
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine (N=995) | 5-Fluorouracil + Leucovorin (N=974)
Diarrhoea (Gastrointestinal disorders) | 437 | 610
Nausea (Gastrointestinal disorders) | 334 | 459
Stomatitis all (Gastrointestinal disorders) | 218 | 574
Vomiting (Gastrointestinal disorders) | 147 | 199
Abdominal pain (Gastrointestinal disorders) | 133 | 149
Constipation (Gastrointestinal disorders) | 86 | 103
Abdominal pain upper (Gastrointestinal disorders) | 70 | 65
Dyspepsia (Gastrointestinal disorders) | 59 | 48
Palmar-plantar (Skin and subcutaneous tissue disorders) | 593 | 85
Erythrodysaesthesia syndrome Alopecia (Skin and subcutaneous tissue disorders) | 63 | 218
Rash (Skin and subcutaneous tissue disorders) | 70 | 80
Erythema (Skin and subcutaneous tissue disorders) | 58 | 51
Fatigue (General disorders) | 155 | 150 — General Disorders and Administration Site Conditions
Asthenia (General disorders) | 96 | 95 — General Disorders And Administration Site Conditions
Lethargy (General disorders) | 97 | 92 — General Disorders And Administration Site Conditions
Pyrexia (General disorders) | 68 | 78 — General Disorders And Administration Site Conditions
Dysgeusia (Nervous system disorders) | 59 | 89
Headache (Nervous system disorders) | 51 | 59
Anorexia (Metabolism and nutrition disorders) | 90 | 104
Conjunctivitis (Eye disorders) | 47 | 60
Dizziness (Nervous system disorders) | 62 | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.